CLINICAL TRIAL: NCT04819178
Title: Real Life Evaluation of SGLT2 Use in Type 1 Diabetes
Acronym: RESGUE1
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawel of approvement of Dapagliflozin to type 1 diabetes
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Peter Rossing, Professor, DM, Peter Rossing, Steno Diabetes Center Copenhagen
Other Study IDs: 22436292
Record Dates: First submitted 2021-03-15; First posted 2021-03-26 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetic Ketoacidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary aim of the study is to prospectively monitor the risk of diabetic ketoacidosis (DKA) during treatment with sodium-glucose cotransporter 2 (SGLT2) inhibitors in type 1 diabetes after the treatment has become available as an adjunct therapy for people with type 1 diabetes.

DETAILED DESCRIPTION:
SGLT2 inhibitors have recently been approved for treatment of type 1 diabetes. SGLT2 inhibitors affect renal glucose transport and promotes glucose excretion in the urine. This have attractive effects, notably by lowering of blood glucose without any increased risk of hypoglycemia as well as a reduction in body weight. Since the risk of hypoglycemia and weight gain during intensification of insulin treatment is a significant barrier for optimal glycemic control, SGLT2 inhibitors could be an attractive adjunct therapy in type 1 diabetes. Furthermore, SGLT2 inhibitors have beneficial cardiovascular and renal effects in persons with type 2 diabetes. This may also benefit persons with type 1 diabetes. However, the major limitation for an universal use of SGLT2 inhibitors in type 1 diabetes is a substantial increase in ketogenesis and the risk of DKA. DKA remain a substantial cause of morbidity and mortality in persons with type 1 diabetes.

Since no data exist on the risk of DKA during SGLT2 inhibition outside the randomized controlled trials, the investigators will initiate a nationwide monitoring study on the use of SGLT2 inhibitors in type 1 diabetes. This will ensure follow-up on the efficacy, safety and patient-reported outcome measures for SGLT2 inhibitors treatment of type 1 diabetes in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* All patiens with type 1 diabetes on SGLT2 inhibitor treatment or where this treatment is planned.

Exclusion Criteria:

* None

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with type 1 diabetes initiated on SGLT2 inhibition will be prospectively included after provision of informed consent. We have established a national network of centers and investigators involved in the treatment of type 1 diabetes. We aim to offer inclusion in the study to every individual where SGLT2 inhibitor treatment is planned
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Diabetic ketoacidosis | 3 years
  Registration of incidents of DKA will be done based on data from medical records, as well as reporting from patients and registries.

SECONDARY OUTCOMES:
Efficacy of treatment | 3 years
  Data on HbA1c and total daily insulin dose will be registered from medical journals at baseline and each year at follow-up together with information on whether patients are still treated with SGLT2 inhibitors. Data on weight and hypoglycemia are obtained from patients.
Patient reported outcome | 3 years
  Patients will be asked to complete the questionnaire "PAID20" (Problem Areas In Diabetes), lowest score is 0, highest score is 80. The higher score the more emotionel reactions the person with type 1 diabetes has. The second questionaire is concernig incidense of being admittet to the hospital with ketoacidosis or hypoglycemia, whether the person with type 1 diabetes has expirienced side effects or weight loss efter initiation of treatment.
Side effects | 3 years
  Registration of incidence of urogenital infection will be done based on data from medical records, as well as reporting from patients and registries.
Hypoglyceamia | 3 years
  Registration of incidence of hypoglycemia will be done based on data from medical records, as well as reporting from patients and registries.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Persson, MD, DMsc, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (3):
- Denmark (3):
  - Steno Diabetes Center Aarhus, Aarhus
  - Steno Diabetes Center Copenhagen, Gentofte Municipality
  - Steno Diabetes Center Region Sjaelland, Køge